CLINICAL TRIAL: NCT00700232
Title: Mutations and Polymorphisms of Gene ABCB4 Among Women Suffering From Intrahepatic Cholestasis of Pregnancy. A Study With a Control Group.
Brief Title: ABCB4 Gene Mutations in Intrahepatic Cholestasis of Pregnancy and Controls
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours, University Hospital, Tours
Other Study IDs: AOHP06-YB GEN CIG
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: genetics; gene expression; MDR3; estrogens; cholestasis; pregnancy; controls
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Normal multiparous pregnant women without intrahepatic cholestasis of pregnancy (control group)

SUMMARY:
Mutations of the ATP binding cassette subfamily B member 4 (ABCB4) gene, a gene involved in a subtype of progressive familial intrahepatic cholestasis, have been reported in women suffering from intrahepatic cholestasis of pregnancy. The true incidence and the role of these ABCB4 gene mutations in patients suffering from intrahepatic cholestasis of pregnancy have not been clearly established.

The aim of the present study is to describe the nature and frequency of these mutations in a series of patients with intrahepatic cholestasis of pregnancy and to compare with a control group of pregnant women without intrahepatic cholestasis of pregnancy.

DETAILED DESCRIPTION:
Intrahepatic cholestasis of pregnancy was defined by pruritus and elevated serum alanine aminotransferase activity or bile acid concentration, with recovery after delivery. Patients with intercurrent liver disease were excluded.

The entire ABCB4 gene coding sequence and the promoter region were analyzed, during the routine medical management, by single strand conformation polymorphism and/or sequencing in 50 unrelated Caucasian patients with intrahepatic cholestasis of pregnancy.

The genomic variants detected in these patients with intrahepatic cholestasis of pregnancy will be sought in 100 control women from Caucasian origin recruited in the same hospital.

ELIGIBILITY:
For the control group :

Inclusion Criteria:

* pregnant woman (age > 18 years) during the third trimester
* caucasian and born in France
* multiparous (with at least 2 full term pregnancies)
* with informed written consent

Exclusion Criteria:

* generalized pruritus and/or liver disease during pregnancy
* liver disease secondary to oral contraception
* Chronic liver disease
* disease during current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: multiparous normal pregnant women (control group)from a single University center
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BACQ Yannick, MD, Study Director — Service d'hépato-gastro-entérologie CHRU Tours
Locations (1):
- Service de Gynécologie Obstétrique CHRU Tours, Tours, France